CLINICAL TRIAL: NCT03869606
Title: A Trial of a Non-Invasive Cardiac Output Monitor to Determine Fluid Responsiveness in Children
Brief Title: Non-Invasive Cardiac Output Monitor in Children
Acronym: NICOM2
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Stasic, Associate Professor of Anesthesia, Indiana University
Other Study IDs: 1808715198
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Output, Low; Pediatric
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: NICOM by Cheetah Medical — Observational measurement, Cardiac Output, Pre- and Post Anesthesia

SUMMARY:
This study will be the first of several studies that establish the value of measuring fluid responsiveness in children undergoing general anesthesia. The first study in this series will determine whether fluid responsiveness, as measured with the NICOM cardiac output monitor in normal children before and after passive leg raising, predicts changes in stroke volume, cardiac output, and blood pressure during the early stages of anesthesia. A second study will determine if early treatment of the fluid responsiveness will prevent the decline in blood pressure that accompanies general anesthesia. If the NICOM monitor permits accurate prediction in normal patients, future studies of pediatric patients undergoing major surgery would be indicated.

The investigators would like to add 25 additional patients who will have the NICOM assessments performed in the pre operative area - Pre anesthesia. General anesthesia may alter the results of the NICOM assessments. The investigators will use these 25 subjects to serve as a comparison/control group.

DETAILED DESCRIPTION:
Eligible patients will be identified from the surgery schedule and will be contacted by a research team member via phone ahead of their surgery date to inform them of the research study. This call will allow the research team member to answer questions and establish the subject's interest in participation. If interested, or not able to be contacted by phone, patient/family will be approached in the pre-operative area or other private hospital setting. He/she and their parent(s) will have ample time to read the consent and ask any questions regarding the study.

If the subject and his/her parent(s) agree to participate, all standard techniques for general anesthesia compatible with the particular surgical procedure will be employed. Clinical decisions concerning the subject's perioperative care will be made by the anesthesiologist of record.

Cardiac output will be measured with the NICOM cardiac output monitor. The NICOM is a non-invasive monitor using bioreactance, a proprietary technique developed by Cheetah Medical that utilizes delay time shifts to measure stroke volume when an alternating current is passed through the thorax. It requires the placement of four surface electrodes (similar to ECG electrodes) above and below the heart on each side of the patient's chest.

This study will measure cardiac output, stroke volume, and fluid responsiveness (increase in stroke volume > 10%) obtained via passive leg elevation immediately after induction of anesthesia. Adult studies have demonstrated that fifty percent of fasted patients are fluid responsive. The investigators seek to determine the incidence on children.

All decisions concerning clinical care of the subject during the perioperative period will made by the anesthesiologist of record in accordance with accepted standard of care.

1. The NICOM® electrodes will be applied in proper position in the pre-op area. In pre-op, baseline and passive leg measurements will be recorded using the NICOM®. Electrodes will remain in place and will again be used during the OR NICOM® measurements.
2. Standard physiologic monitors will be used: non-invasive blood pressure, ECG, pulse oximeter, capnograph (end-tidal carbon dioxide), BIS (bispectral analsysis/depth of anesthesia).
3. Induction of anesthesia to be determined by the anesthesiologist of record. May be either inhalation or intravenous.
4. Measurements recorded after application of NICOM electrodes include blood pressure, heart rate, end-tidal carbon dioxide, arterial oxygen saturation, BIS level, stroke volume, cardiac output.
5. After measurement of baseline cardiorespiratory parameters, passive leg elevation to 45 degrees will be performed.
6. Cardiorespiratory measurements describe in section d will be repeated after passive leg elevation.
7. Cardiorespiratory parameters will be measured during the next 60 minutes of anesthesia. This information will be used to determine whether fluid responsive patients require additional intravenous fluids or vasoactive drugs during the course of anesthesia.

The same procedures listed above will be performed Pre-anesthesia in the Pre operative area, while the subject is fully awake.

General anesthesia may alter the results of the NICOM procedures. The investigators will add 25 patients who will be evaluated with the study procedures pre anesthesia as a control/comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 11 to no older than 17 years of age

Exclusion Criteria:

* severed developmental delay,
* orthopedic patients with leg injuries
* injury that would prevent passive leg elevation.
* severe aortic insufficiency,
* severe anatomic abnormalities of the thoracic aorta
* patients with external cardiac pacemakers. close

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy 10 to 17 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Output via NICOM monitor | Pre-Induction and fifteen minutes up to thirty minutes Post-Anesthesia Induction
  Stroke volume x Heart Rate = Cardiac Output

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F Stasic, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No